CLINICAL TRIAL: NCT04394312
Title: Parent PLAYSHOP: A Physical Literacy Training Workshop for Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Victoria (Other)
Responsible Party: Principal Investigator, Valerie Carson, Associate Professor, University of Alberta
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PLAYSHOP
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Motor Activity; Parent-Child Relations
Keywords: Questionnaires; Interviews, Telephone
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants are assigned to the intervention group or control group.
Masking Description: As this was a pragmatic intervention participants, investigators, and outcome assessors were aware of the group allocation based on the workshop they attended and the survey data collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will attended a 75 minute physical literacy workshop (Parent PLAYSHOP). A questionnaire will be completed at the beginning of the workshop and the end of the workshop to measure if there is a difference in parent's knowledge and confidence levels in regard to engaging in meaningful physical activity with their children.
  Interventions: Other: Parent PLAYSHOP
- Control (No Intervention): Participants will complete the 2 questionnaires online, one week or more apart. Once questionnaires are completed they will be invited to attended the 75 minute physical literacy workshop. The workshop content and delivery will be the same as the intervention group but will not include questionnaires.

INTERVENTIONS:
Other: Parent PLAYSHOP — The Parent PLAYSHOP includes:
  1. Educational Training- the 75 min workshop will be delivered by a trained facilitator. Parents will be introduced to physical literacy via education, group discussion, and active participation in fundamental movement skills (FMS) based activities. Parents will be provided with modifications to perform activities 'at home'.
  2. Distribution Education and Activity Resources- At the workshop conclusion parents are given education Resources (e.g. Canada's 24-hour movement guidelines for the early years, activity idea booklet, and a physical literacy handout) and inexpensive activity resources (ball, bean bag, scarves, balloons etc.).
  3. Provide Follow-up Support- Research staff will send parents a follow-up email with key workshop messages (e.g., rationale and importance of physical literacy); support and encouragement for parents to engage in purposeful play with their child; and an opportunity for parents to provide feedback and/or seek further support.
  Arms: Intervention

SUMMARY:
The objective of this research is to 1) determine the impact of a physical literacy training workshop for parents of preschool children (3-5 years) on their knowledge and confidence levels in regards to engaging in meaningful physical activity with their child(ren) in order to promote physical literacy. 2) Evaluate workshop reach and implementation facilitators and barriers.

In this pilot study, interested participants will be randomized into the intervention group or the wait-list control group. Participants will complete two brief surveys regarding their knowledge and confidence in doing physically activities with their children. The intervention group will receive a 75 minute physical literacy workshop at baseline, and complete a 2 month follow-up interview. The wait-list control group will receive the workshop after questionnaires have been completed.

Statistical analysis will be conducted to compare change in knowledge and confidence levels in between intervention and control groups. Findings will contribute to promoting and improving parental confidence in providing opportunities for children to develop their physical literacy and advance future research regarding physical activity promotion for children.

DETAILED DESCRIPTION:
Purpose/objective: 1)Determine if a physical literacy training workshop can increase parental knowledge, confidence levels, and improve parenting practices related to engaging in play with their preschool child(ren) that facilitates the development of physical literacy. 2) Evaluate workshop reach and implementation facilitators and barriers.

Hypothesis: 1)Parents in the intervention group will have a larger increase in parental knowledge and confidence levels in regards to engaging in meaningful play with their preschool child(ren) than parents in the control group. 2) Parents will report satisfaction with the implementation and that they changed parenting practices related to physical activity at the 2 month follow-up.

Justification: Preschoolers are typically at a development stage where they are beginning to possess a unique set of motor skills that allow them to engage in a wider range of physical activities. Parents have been identified as a key gatekeeper for physical activity in children.

Research method: This pilot study is a Type 1 Hybrid Effectiveness Trial, where an intervention is tested while also gathering information on the effectiveness and potential for real world use (Curran et al., 2012). Approximately, 100 participants will be randomized into an intervention group or a wait-list control group across two Canadian data collection sites: Edmonton, Alberta and Victoria, British Columbia. Participants in the intervention group will receive a 75 minute physical literacy workshop in their community (e.g. community recreation centre, local school, family resource centre) at baseline, where their preschool child is encouraged to attend and participate. The workshop will provide parents with physical literacy training including modifications for the home setting.The overall aim of the workshop is to support parents in engaging in play with their child that facilitates the development of physical literacy. The program was designed using Bandura's social cognitive theory (Bandura, 1986) with a specific emphasis on parent's self-efficacy and related intervention change techniques described using the Behavior Change Wheel (BCW; a synthesis of 19 behavior change frameworks). To address the 1st objective, the intervention group will complete a brief pre-workshop questionnaire, post-workshop questionnaire, and a follow-up interview approximately 2 months after the workshop. At the end of the workshop, parents will take home a goody bag with basic and inexpensive play equipment/resources. In between the workshop and the 2 month follow-up, they will receive at least two booster e-mails/texts with play ideas. The wait-list control group will complete the two questionnaires online (approximately 1 week apart) around the same time as the intervention group and receive the workshop at a later date. The control group will also receive the goody bag. To address the 2nd objective, parents will report their satisfaction and facilitators and barriers to implementing activities and research staff/partners that delivered the workshops will be invited to be interviewed at the end of the study in order to evaluate reach and implementation facilitators and barriers .

Plan for data analysis: Repeated measures ANOVA and/or linear mixed models will be used to compare change in knowledge and confidence levels between intervention and wait-list control groups (Objective 1). Thematic analysis will be used to analyze parent's satisfaction and changes in parenting practices reported in the 2 month follow-up interview (Objective 1). Thematic analysis will also be used to evaluate the reach and implementation facilitators and barriers reported by parents and research staff/partners (Objective 2).

ELIGIBILITY:
Inclusion Criteria:

* Parents with a pre-school aged child (3-5 years old)

Exclusion Criteria:

* Parents that are not comfortable speaking and reading English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in parental knowledge, confidence, and intention in engaging in purposeful play with their preschool child(ren) that builds physical literacy. | Before and immediately after the 75 minute workshop
  The pre and post workshop questionnaires will assess changes in parent's knowledge and confidence of specific physical literacy components (e.g. manipulative skills, locomotor skills, balance and stability skills) and intention to engage in purposeful play with their preschool child(ren).
Changes in parenting practices regarding engagement in purposeful play. | Approximately 2 months after attending the workshop
  In the semi- structured interview approximately 2 months after the PLAYSHOP, parents will be asked about changes in their parenting practice regarding engagement in meaningful activities with their preschool child(ren) that builds physical literacy.

SECONDARY OUTCOMES:
Parental satisfaction and implementation barriers and facilitators. | Approximately 2 months after attending the workshop
  In the semi- structured interview approximately 2 months after the PLAYSHOP, parents will report their satisfaction with the workshop. Parents will also be asked what facilitators and barriers they have experienced while implementing physical literacy activities in their home since the workshop.
Intervention reach and workshop implementation barriers and facilitators. | After study completion, approximately 6 months from start of project
  In the semi-structured interview with research staff/partners, participants will report facilitators and barriers of workshop delivery and proposed changes.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie L Carson, PhD, Principal Investigator — University of Alberta; Patti-Jean Naylor, PhD, Principal Investigator — University of Victoria
Locations (2):
- Canada (2):
  - University of Alberta, Van Vliet Complex, Edmonton, Alberta
  - University of Victoria, McKinnon Building, Victoria, British Columbia

IPD SHARING:
Plan to Share IPD: No
To protect participant's personal data IPD will not be shared with other researchers.

REFERENCES:
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Bandura A. Social foundations of thought and action. Englewood Cliffs, NJ, 1986.
- [Derived] Lane C, Naylor PJ, Predy M, Kurtzhals M, Rhodes RE, Morton K, Hunter S, Carson V. Exploring a parent-focused physical literacy intervention for early childhood: a pragmatic controlled trial of the PLAYshop. BMC Public Health. 2022 Apr 5;22(1):659. doi: 10.1186/s12889-022-13048-5. PMID 35382793